CLINICAL TRIAL: NCT04634370
Title: Fase I Clinical Trial on Natural Killer Cells for COVID-19
Brief Title: Fase I Clinical Trial on NK Cells for COVID-19
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20200210
Record Dates: First submitted 2020-11-16; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Covid19; Sars-cov 2
Keywords: Natural Killer Cells; COVID-19; Sars-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Each patient will receive on dose of intravenous natural killer cell in following levels:
  Level 1 : 1x106 cells/kg body weight (patients 1 to 3) Level 2: 5x106 cells/kg body weight (patients 4 to 6) Level 3: 1x107 cells/kg body weight (patients 7 to 24)
  Interventions: Biological: Natural Killer Cells infusion

INTERVENTIONS:
Biological: Natural Killer Cells infusion — Each patient will receive on dose of intravenous natural killer cell in following levels:
  Level 1 : 1x106 cells/kg body weight (patients 1 to 3) Level 2: 5x106 cells/kg body weight (patients 4 to 6) Level 3: 1x107 cells/kg body weight (patients 7 to 24)

SUMMARY:
Coronavirus Disease 2019 (COVID-19) is spreading worldwide and has become a public health emergency of major international concern. Currently, no specific drugs or vaccines are available.

This study aims to investigate the safety and efficacy of intravenous infusion of natural killer cells patients with COVID-19.

DETAILED DESCRIPTION:
In March 2020, the World Health Organization secreted COVID-19 as a pandemic. Although most infected individuals can develop effective immunity, the population at risk (elderly, obese and individual with comorbidities) develop a rapid and frequently fatal disease, with severe acute respiratory syndrome, cytokine storm and coagulopathies; for those who recover, severe pulmonary sequels are frequently observed. We propose a phase I clinical trial to test safety and feasibility of NK cells adoptive immunotherapy for COVID-19. Natural Killer cells are innate granular lymphocytes able to rapidly recognize and kill, without previous exposition, altered cells; it is widely recognized as immune effectors specialized in lysing virus infected cells releasing antigens and activating cytokines to antigen presenting cells and, by doing so, stimulating effective adaptive immunity. We hypothesize that the early infusion of highly activated NK cells will activate adaptive immune effectors preventing the severe clinical evolution of COVID-19 infection. Adoptive NK cell immunotherapy for severe virus infections is innovative. Our proposition is in line with the Brazilian Public Health system purposes, which is to offer secure and effective therapies for all COVID-19 infected individuals. Upon proving NK cell immunotherapy effectiveness for serious virus infections, we can evolve to test this strategy for common viruses that cause epidemics and endemics such as the ones caused by Dengue, Zika, Chikungunya, C and B hepatitis and HIV.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmation of COVID19 infection by reverse-transcription polymerase chain reaction (RT-PCR);
* The patient or legal donor agrees to participate in the study and signs the informed consent;
* Patients with white or yellow criteria according to the score proposed by Liao et al (2020).

Exclusion Criteria:

* Patient with pregnancy, are planning to become pregnant or breastfeeding;
* Patients with malignant blood-borne diseases such as HIV or syphilis;
* Not consenting for clinical trial;
* Patients with other than white or yellow criteria according to the score proposed by Liao et al (2020).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-01-02 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 30 days
  Assessment of Overall survival at 30 days post intervention
Changes on inflammatory C-reactive protein | 60 days
  To assess the anti-inflammatory effect of the proposed treatment with assessment of the levels of C-reactive protein (mg/dL)
Hospital stay | 60 days
  days of the patients in hospital
Oxygenation index (PaO2/FiO2) | 60 days
  Evaluation of functional respiratory changes: PaO2 / FiO2 ratio
Improvement in Liao's score (2020) | 60 days
  Improvement in Liao's score (2020)
Radiological improvement | 60 days
  Computed tomography Chest assesment will be done to assess improvement in radiological findings of COVID-19

CONTACTS AND LOCATIONS:
Overall Officials: Lucia Silla, MD, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No